CLINICAL TRIAL: NCT04359680
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Pre- and Post Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses (VRI) in Healthcare Workers and Others at Increased Risk of SARS-CoV-2 Infection
Brief Title: Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Pre- and Post Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses (VRI) in Healthcare Workers and Others at Increased Risk of SARS-CoV-2 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RM08-3007
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Viral Respiratory Illnesses
Keywords: COVID-19; Viral Respiratory Illnesses
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two NTZ 300 mg tablets orally twice daily for 6 weeks.
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super B-Complex
- Placebo (Placebo Comparator): Two placebo tablets orally twice daily for 6 weeks.
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin Super B-Complex

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 600 mg administered orally twice daily for six weeks
  Other Names: NTZ (nitazoxanide); NT-300
  Arms: Nitazoxanide
Drug: Placebo — Placebo administered orally twice daily for six weeks
  Arms: Placebo
Dietary Supplement: Vitamin Super B-Complex — Vitamin Super B-Complex administered orally twice daily to maintain the blind

SUMMARY:
Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Pre- and Post Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses (VRI) in Healthcare Workers and Others at Increased Risk of SARS-CoV-2 Infection

DETAILED DESCRIPTION:
Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Pre- and Post Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses (VRI) in Healthcare Workers and Others at Increased Risk of SARS-CoV-2 Infection

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age or of legal consenting age based on local requirements.
2. Persons at increased risk of contracting COVID-19, including:

   1. Healthcare workers with known direct occupational exposure to COVID-19 within 7 days prior to enrollment. A qualifying person (i) provides healthcare to patients and/or (ii) typically positions themselves within 6 feet of patients ("close contact") and (iii) is a full- time employee (average of ≥ 24 hours/week) in a high contact area (Emergency Department, Intensive Care Unit, COVID-specific Care Unit, Walk-in Clinic, Paramedic/First Responder).
   2. Persons participating in social activities without the practice of generally accepted social distancing practices at least three times per week. Qualifying activities include the presence of at least 10 people in close (<6 feet) proximity to each other without masks or other personal protective equipment (e.g., socializing at bars or community/social centers, in-home social gatherings, classes or trainings, etc.). These subjects must have engaged in such activities at least three times in the past 7 days and plan to continue these activities during the study.
3. Must have a smartphone, tablet, computer, or other qualifying internet- enabled device and daily internet access.
4. Occupational exposure to a person infected with SAR-CoV-2 within 7 days prior to enrollment or social interaction as defined in criterion 2(b).
5. Willing and able to provide written informed consent and comply with the requirements of the protocol, including completion of the subject diary.

Exclusion Criteria:

1. Subjects not at increased risk of contracting SARS-CoV-2 from occupational or social behaviors.
2. Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
3. Subjects with a history of COVID-19 or known to have developed anti- SARS-CoV-2 antibodies or received a SARS-CoV-2 vaccine.
4. Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions or antiviral therapy for influenza within two weeks prior to and including study day 1.
5. Subjects residing in the same household with another family member currently participating in the study.
6. Receipt of any dose of NTZ within 7 days prior to screening.
7. Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
8. Known sensitivity to NTZ or any of the excipients comprising the study medication.
9. Subjects unable to swallow oral tablets or capsules.
10. Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycle prior to study drug administration, an (intrauterine device) IUD, or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
11. Females who are breastfeeding.
12. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
13. Subjects taking medications considered to be major CYP2C8 substrates.
14. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1407 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - HealthStar Research LLC, Hot Springs, Arkansas
  - So Cal Clinical Research, Huntington Beach, California
  - Long Beach Clinical Trials, LLC, Long Beach, California
  - Meris Clinical Research, Brandon, Florida
  - Invesclinica US LLC, Fort Lauderdale, Florida
  - The Chappel Group Research, Kissimmee, Florida
  - New Horizon Research Center, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - DMI Research, Pinellas Park, Florida
  - Tampa General Hospital, Tampa, Florida
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Chicago Medical Research Institute, Inc., Chicago, Illinois
  - Quad Clinical Research, Chicago, Illinois
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Vida Clinical Studies, Dearborn, Michigan
  - Beacom Family Health Connection, Fremont, Nebraska
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - The New York Center for Travel and Tropical Medicine, New York, New York
  - RH Medical Urgent Care Professional PLLC, The Bronx, New York
  - Centex Studies, Inc., Houston, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - LinQ Research LLC, Pearland, Texas
  - Rio Grande Valley Clinical Research Institute, Pharr, Texas
  - BFHC Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 711 | 696
Completed | 616 | 604
Not Completed | 95 | 92
Not completed — Withdrawal by Subject | 29 | 24
Not completed — Adverse Event | 6 | 2
Not completed — Lost to Follow-up | 56 | 59
Not completed — Protocol Violation | 3 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population consists of all subjects receiving at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 686 | 663 | 1349
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13.8) | 40 (13.8) | 40 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 410 | 411 | 821
  Male | 276 | 252 | 528
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 219 | 219 | 438
  Not Hispanic or Latino | 455 | 429 | 884
  Unknown or Not Reported | 12 | 15 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 6
  Asian | 33 | 25 | 58
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 118 | 123 | 241
  White | 469 | 469 | 938
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 56 | 45 | 101
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 84 (22.4) | 85 (22.1) | 84 (22.2)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Symptomatic Laboratory-confirmed COVID-19 Identified After Start of Treatment and Before the End of the 6-week Treatment Period.
Time Frame: Up to 6 weeks
Population: The intent-to-treat (ITT) population consists of all subjects who received at least one dose of study medication and were negative for all respiratory viruses tested at Baseline. Proportions were rounded to the nearest hundredth decimal.
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 629 | 613
proportion of participants | 0.02 | 0.02
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.9434, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.0290, 95% CI 2-sided [0.4696 to 2.2546]

2. Primary Outcome: The Proportion of Subjects With Symptomatic Laboratory-confirmed VRI Identified After the Start of Treatment and Before the End of the 6-week Treatment Period.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 629 | 613
proportion of participants | 0.05 | 0.05
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.6805, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.1162, 95% CI 2-sided [0.6623 to 1.8813]

3. Secondary Outcome: Proportion Experiencing Mortality Due to COVID-19 or Complications Thereof
Description: Note: statistical analysis not performed because no events occurred.
Time Frame: Up to 8 weeks
Population: The intent-to-treat (ITT) population consists of all subjects who received at least one dose of study medication and were negative for all respiratory viruses tested at Baseline
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 629 | 613
proportion of participants | 0 | 0

4. Secondary Outcome: Proportion With Anti-SARS-CoV-2 Antibodies at Either of the Week 6 or Week 8 Visits
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 629 | 613
proportion of participants | 0.17 | 0.19
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.3459, Cochran-Mantel-Haenszel

5. Post Hoc Outcome: Days Not at Usual Health Due to COVID-19
Description: Descriptive statistics of the number of days patients with symptomatic COVID-19 report not being at usual health due to COVID-19
Time Frame: Up to 56 days
Population: Participants experiencing symptomatic COVID-19 during the study period
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 13 | 13
days | 13.2 (16.88) | 19.5 (14.58)

6. Post Hoc Outcome: Days Unable to Perform Usual Activities Due to COVID-19
Description: Descriptive statistics of the number of days patients with symptomatic COVID-19 report being unable to perform usual activities due to COVID-19
Time Frame: Up to 56 days
Population: Patients with symptomatic COVID-19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 13 | 13
days | 8.2 (11.73) | 16.5 (12.72)

7. Post Hoc Outcome: Days Meeting Acute Respiratory Illness Symptom Severity Criteria Due to COVID-19
Description: Descriptive statistics of the number of days patients with symptomatic COVID-19 met the protocol-specified acute respiratory illness symptom severity criteria due to COVID-19
Time Frame: Up to 56 days
Population: Patients with symptomatic COVID-19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 13 | 13
days | 10.0 (15.52) | 13.8 (12.05)

8. Post Hoc Outcome: Maximum Symptom Severity Due to COVID-19
Description: Descriptive statistics of the maximum symptom severity reported by patients with symptomatic COVID-19. The global assessment of symptom severity was reported by patients as "absent", "mild", "moderate", "severe", or "very severe" and coded as 0, 1, 2, 3, or 4, respectively.
Time Frame: Up to 56 days
Population: Participants with symptomatic COVID-19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale | 1.3 (0.95) | 2.3 (1.11)

9. Post Hoc Outcome: Days Not At Usual Health Due to VRI
Description: Descriptive statistics of the number of days patients with symptomatic viral respiratory illness (VRI) report not being at usual health due to VRI
Time Frame: Up to 56 days
Population: Participants experiencing symptomatic viral respiratory illness
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 29 | 31
days | 9.9 (12.19) | 14.4 (14.44)

10. Post Hoc Outcome: Days Unable to Perform Usual Activities Due to VRI
Description: Descriptive statistics of the number of days patients with symptomatic viral respiratory illness (VRI) report being unable to perform usual activities due to VRI
Time Frame: Up to 56 days
Population: Participants experiencing symptomatic viral respiratory illness (VRI)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 29 | 31
days | 5.9 (8.85) | 9.7 (11.61)

11. Post Hoc Outcome: Days Meeting Acute Respiratory Illness Symptom Severity Criteria Due to VRI
Description: Descriptive statistics of the number of days patients with symptomatic viral respiratory illness (VRI) met the protocol-specified acute respiratory illness symptom severity criteria due to VRI
Time Frame: Up to 56 days
Population: Participants with symptomatic viral respiratory illness (VRI)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 29 | 31
days | 7.3 (10.97) | 11.4 (12.73)

12. Post Hoc Outcome: Maximum Symptom Severity Due to VRI
Description: Descriptive statistics of the maximum symptom severity reported by patients with symptomatic viral respiratory illness (VRI). The global assessment of symptom severity was reported by patients as "absent", "mild", "moderate", "severe", or "very severe" and coded as 0, 1, 2, 3, or 4, respectively.
Time Frame: Up to 56 days
Population: Participants with symptomatic viral respiratory illness (VRI)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 29 | 31
score on a scale | 1.6 (0.98) | 1.9 (1.01)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/686 | 0/663
Serious Adverse Events (participants affected / at risk) | 3/686 | 6/663
Other Adverse Events (participants affected / at risk) | 0/686 | 0/663
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=686) | Placebo (N=663)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04359680/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04359680/SAP_001.pdf